CLINICAL TRIAL: NCT01488357
Title: Patient Preferences for Breast Reconstruction After Mastectomy
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); North Carolina TraCS Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: 11-0119; 1K07CA154850-01A1 (NIH)
Record Dates: First submitted 2011-10-12; First posted 2011-12-08 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; UNC; Lineberger; Breast Reconstruction; Mastectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Early stage breast cancer patients receiving mastectomy

SUMMARY:
Deciding whether or not to have breast reconstruction after mastectomy is highly challenging for many patients. This study will examine patients' decisions about reconstruction and the effects of reconstruction on quality of life and body image.

DETAILED DESCRIPTION:
Breast reconstruction after mastectomy is an important treatment option for the many thousands of women who undergo mastectomy each year. Its insurance coverage is mandated by federal law. Many women who want reconstruction, particularly women from racial and ethnic minorities, never receive it, and some women who undergo reconstruction regret having it, raising concern about the quality of decisions about the procedure. Little is known about the quality of breast reconstruction decisions, defined as the extent to which decisions are informed and concordant with patients' preferences. A lack of reliable methods for evaluating preference concordance has resulted in a paucity of research in this area. Deciding about breast reconstruction requires a patient to predict how she would feel after the procedure, a process called affective forecasting. Extensive psychological research has shown that people have difficulty making accurate predictions about how they will feel, tending to overestimate the effects of disease and treatments on their well-being and to underestimate their ability to adapt to change and the effects of other aspects of their lives. Despite the importance of affective forecasting to decisions about breast reconstruction, no research has examined this aspect of those decisions. The investigator proposes to conduct a pilot cohort study of breast cancer patients undergoing mastectomy, with or without reconstruction with the following specific aims: Aim 1: to evaluate whether patients make informed decisions about breast reconstruction that are concordant with their preferences; Aim 2: to assess the accuracy of patients' preoperative predictions about their post-operative body image and well-being; and Aim 3: to assess the effects of breast reconstruction on quality of life and body image and the potential modification of those effects by preference concordance.

ELIGIBILITY:
Inclusion Criteria:

* Women 21 years of age or older
* Having a mastectomy at UNC for treatment of Stage I, II, or III breast cancer, ductal carcinoma in situ (DCIS) or for prophylaxis

Exclusion Criteria:

* Stage IV breast cancer
* Women who do not speak English
* Severe psychiatric illness

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women undergoing mastectomy at UNC for treatment of Stage I, II, or III breast cancer or DCIS, or for prophylaxis
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02-27 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Treatment Concordance | Time of Surgery decision which is an average of 2-4 weeks before surgery.
  The investigator will assess patient preferences pre-operatively using conjoint analysis. The investigator will determine if these preferences are concordant with the patient's treatment decision.

SECONDARY OUTCOMES:
Body Image | 18 months post operatively
  Body Image Scale
Satisfaction with Decisions | 18 months post-operatively
  Satisfaction with Decisions Scale
Quality of Life | 18 months post-operatively
  Breast-Q and Forecasting measures
Knowledge | Pre-operatively at time of decision making which is an average of 2-4 weeks before surgery.
  The investigator will use the Decision Quality Instrument which includes knowledge questions to assess patient understanding of breast reconstruction.

CONTACTS AND LOCATIONS:
Overall Officials: Clara N Lee, MD, MPP, Principal Investigator — Ohio State University
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: National Cancer Institute — http://www.cancer.gov/
- See also: UNC Lineberger Comprehensive Cancer Center — http://cancer.unc.edu/